CLINICAL TRIAL: NCT03199196
Title: Using Social Networks to Promote Physical Activity in African American and Hispanic Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-0717
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Cancer Prevention
Keywords: Cancer Prevention; African-American woman; Hispanic woman; Sedentary; Activity Tracker; Smartphone Application; Questionnaires; Surveys; Focus Group; Electronic Newsletters; Telephone Counseling
MeSH Terms: conditions — Sedentary Behavior | interventions — Fitness Trackers; Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Intervention (Experimental): Participants given an activity tracker at the given an accelerometer at each visit. Participants instructed in use of a smartphone application at the baseline visit.
  Participant emailed electronic newsletters to read that may help participant be more physically active.
  Research staff provides telephone counseling to participant and partner biweekly during weeks 1-8 (weeks 1, 3, 5, and 7), and monthly during weeks 9-16 (weeks 11 and 15).
  Study visits performed 2 times (1 time at the beginning of the study, and 1 time 16 weeks after beginning the study).
  Participants complete questionnaires 1 time at the beginning of the study, 8 weeks after joining the study, and 16 weeks after beginning the study.
  Participants invited to take part in a final focus group sometime after the 16-week visit.
  Interventions: Device: Activity Tracker; Device: Smartphone Application; Behavioral: Questionnaires; Behavioral: Focus Group; Behavioral: Electronic Newsletters; Behavioral: Telephone Counseling
- Group 2 - Control (Other): Participants sent electronic newsletters throughout the study that may help participant be more physically active.
  Study visits performed 2 times (1 time at the beginning of the study, and 1 time 16 weeks after beginning the study).
  Participants complete questionnaires 1 time at the beginning of the study, 8 weeks after joining the study, and 16 weeks after beginning the study.
  Participants invited to take part in a final focus group sometime after the 16-week visit.
  Interventions: Behavioral: Questionnaires; Behavioral: Focus Group; Behavioral: Electronic Newsletters

INTERVENTIONS:
Device: Activity Tracker — Group 1 - Intervention: Participants given an accelerometer at each visit. Participant wears the accelerometer for 7 days.
  Group 2 - Newsletters: After completing the 16 week visit, participant given an activity tracker.
  Arms: Group 1 - Intervention
Device: Smartphone Application — Group 1 - Intervention: Participant given smartphone application baseline visit to track physical activity, connect with participant's partner to share information about participant's physical activity, and provide support to partner to be more physically active.
  Group 2 - Newsletters: After completing the 16 week visit, participant given instruction in the use of a smartphone application.
  Arms: Group 1 - Intervention
Behavioral: Questionnaires — Participants complete questionnaires about feelings, moods, motivation for physical activity, any social support received from others, the neighborhood participant lives in, and other physical activity-related topics. Questionnaires completed 1 time at the beginning of the study, 8 weeks after joining the study, and 16 weeks after beginning the study.The questionnaires should take about 45 minutes to complete.
  Other Names: Surveys
Behavioral: Focus Group — Participants invited to take part in a final focus group. Focus group takes place sometime after the 16-week visit. Focus groups/interviews are audio recorded.
Behavioral: Electronic Newsletters — Participant emailed electronic newsletters to read that may help participant be more physically active.
Behavioral: Telephone Counseling — Research staff provides telephone counseling to participant and partner biweekly during weeks 1-8 (weeks 1, 3, 5, and 7), and monthly during weeks 9-16 (weeks 11 and 15).
  Arms: Group 1 - Intervention

SUMMARY:
The goal of this research study is to learn if enrolling in a program with a partner that involves monitoring each other's physical activity and providing support to one another can help both participants be more physically active.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you and your partner will be randomly assigned (as in a flip of a coin) to be in 1 of 2 groups after you complete the first in-person visit. You will have an equal chance of being in any group.

If you are assigned to Group 1, the following tests and procedures will be performed:

* You will wear an activity tracker that you will be given at the baseline visit. The activity tracker is a small device worn on your wrist that records how many steps you have taken.
* You will be instructed in the use of a smartphone application at the baseline visit which you will use to track your physical activity, connect with your partner to share information about your physical activity, and provide support to your partner to be more physically active.
* You will have 6 counseling calls over the telephone throughout the study with a trained counselor and your partner.
* You will be emailed electronic newsletters to read that may help you be more physically active.

If you are assigned to Group 2, you will be sent the newsletters that may help you be more physically active and upon completing the16 week visit, you will be given an activity tracker and instruction in the use of a smartphone application.

Study Visits:

You will visit MD Anderson Cancer Center, Windsor Village United Methodist Church, or a community site 2 times (1 time at the beginning of the study, and 1 time 16 weeks after you begin the study). Each visit should take about 90 minutes. The following procedures will be performed:

* Your blood pressure will be measured. If you have a blood pressure reading higher than 140/90 mm Hg, you can participate in this study only with a clearance letter from your physician or nurse practitioner. If your blood pressure reading is higher than 180/120 mm Hg, the study staff must contact 911 and have EMS come and treat you due to your blood pressure being dangerously high. You have the right to refuse EMS services but study staff are still required to contact 911 immediately as a precaution. You will not be able to continue in the study until the clearance letter has been received.
* You will complete questionnaires about your feelings, moods, your motivation for physical activity, any social support you may receive from others, the neighborhood you live in, and other physical activity-related topics. The questionnaires should take about 45 minutes to complete. For the 2nd visit, you will have the option of completing the questionnaire online before your scheduled visit. This may reduce the length of your 2nd visit.
* You will be asked about your diet (for example, what you eat and drink each day).
* Your height, weight, and waist and hip circumference will be measured. To measure your waist and hip circumference, you may be asked to lift your shirt to expose your stomach area and lower your pants to expose your mid-hip area. The height, weight, and waist and hip circumference measurements should take about 10 minutes and will be performed in a private area.
* Your heart rate variability (HRV) will be measured with a wrist watch and a belt band. To measure your HRV, you will be asked to lift your shirt to expose your upper stomach area (at the breast bone). The band will be damp and should make firm contact with your skin. °You will wear the device for 5 minutes while it records your HRV as you sit quietly.
* You will be given an accelerometer at each visit. You will wear the accelerometer for 7 days and then return it in an pre-addressed envelope provided to you. An accelerometer is a small device that is worn on your hip that measures the amount of physical activity you do.

At 8 weeks after you begin the study, you will answer some questions either over the phone or through an online survey. The questions will cover the same topics as for the in-person visits. This should take about 30 minutes to complete.

All participants will be invited to take part in a final focus group. This focus group will take place sometime after the 16-week visit. You will be asked what you think about the study, including what you liked, did not like, and how you think it could be improved. If you want to provide this feedback but you cannot come to the focus group, you may provide feedback in another way (such as a phone interview or you could meet the study staff at the church or a community setting). These focus groups/interviews will be audio recorded. Your name and identifying information will be deleted from the recording before being transcribed (typed out) by an outside party. This should take about 90 minutes. The digital audio files will be destroyed within 10 years after publication.

Length of Study:

Your participation on this study will be over after you complete the final focus group visit.

Additional Information:

If you are assigned to Group 1, you may be contacted by phone or mail while you are taking part in this study to remind you about study visits, study procedures, and counseling calls.

You will be asked to give the names and contact information of family members and/or friends for the study staff to contact in the event they cannot reach you first.

The counseling calls for Group 1 will be recorded to monitor counseling procedures.

You will also be asked to participate in two optional procedures. First, you will be asked to "friend" your counselor on the mobile application so that the counselor can monitor your steps in preparation for the counseling calls. Second, you will also be asked to share your user ID and password for the activity tracker. This will enable research staff to download your physical activity data that will help staff to understand how much participants are using the device and how many steps they are taking. These data will only be examined during the 16-week study period, and you will be instructed to change your password at the end of the study.

If the accelerometer is lost or stolen, you will not be responsible for the replacement cost, but you should tell the study staff right away.

You will be able to keep the activity tracker after the study is complete.

Your home address may be used to access public information about the area where you live. This is to help researchers learn about how your neighborhood encourages physical activity. The results from this study will only be reported as a group and you will not be identifiable from any products resulting from this study (such as research papers). Your home address will never be released or published in any form. Your address will be stored separately from other study data, and only the study chair will be able to see the data after the neighborhood information has been collected.

You may be contacted in the future to see if you would agree to take part in other research studies.

Women who are pregnant or thinking about becoming pregnant during the study period will no longer be able to participate. If you become pregnant during this study, please tell the study staff right away.

This is an investigational study.

Up to 64 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported AA race or Hispanic ethnicity (all participants except partners)
2. Age 25-60 years
3. Able to speak English and read at a sixth grade level (as indicated by a score of at least 7 on the Rapid Estimate of Adult Literacy in Medicine, revised [REALM-R]; (Intervention study participants only)
4. Physically able to engage in low-to-moderate PA as assessed by the PA Readiness Questionnaire (PAR-Q), or by physician clearance (Intervention study participants only)
5. Low self-reported moderate-to-vigorous PA (<90 minutes/week)
6. Able to enroll with one female non-spousal family member or friend (Intervention study participants only)
7. Functioning mobile phone capable of accessing the internet and downloading mobile applications ("apps")

Exclusion Criteria:

1. Pregnancy or lactation
2. Participation in the pre-intervention focus groups (Intervention study participants only)
3. Participation in the last 90 days in a research study designed to promote physical activity

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2014-05-02 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Women's Preferences for a Physical Activity (PA) Promotion Intervention | 16 weeks
  Women's preferences for a physical activity (PA) promotion intervention determined by focus groups.

SECONDARY OUTCOMES:
Feasibility of a Social Network-Based Physical Activity (PA) Intervention in Sedentary Women Who are Primarily African American (AA) and Hispanic | 16 weeks
  Study considered feasible only if recruitment and retention percentages reach the lower bound of the one-sided 90% confidence intervals of the target unless there are convincing arguments they can be improved sufficiently by modifying recruitment or retention strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Larkin L. Strong, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Windsor Village United Methodist Church, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org